CLINICAL TRIAL: NCT02248870
Title: Analgesic Duration af a Preoperative Single-shot Femoral Nerve Block With Bupivacaine and Adjuvant Dexamethasone in Patients With Hip Fracture
Brief Title: Femoral Nerve Block With Bupivacaine and Adjuvant Dexamethasone in Patients With Hip Fracture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Less inclusions than expected with the given criteria
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol1tdn
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-03

CONDITIONS: Hip Fracture
Keywords: femoral neck
MeSH Terms: conditions — Hip Fractures | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Bupivacaine with adrenaline with 2 ml. of Saline added
  Interventions: Drug: Saline
- Dexamethasone (Experimental): Bupivacaine with adrenaline with 2 ml. of Dexamethasone added
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone is added to Bupivacaine with Adrenaline for perineural injection
  Arms: Dexamethasone
Drug: Saline — Saline is added as a placebo to Bupivacaine with adrenaline for perineural injection
  Other Names: Solution of sodium chloride
  Arms: Saline

SUMMARY:
Prolongation of the analgesic effect of a femoral nerve block from the present 15 hours to 24 hours in patients with hip fracture would have a major impact in order to provide better preoperative analgesia for this group.

In other trials concerning other nerves then the femoral nerve the addition of Dexamethasone to the local anesthetics doubled the analgesic duration. No studies has investigated the effect of the addition of Dexamethasone to the femoral nerve block in patients with hip fracture.

The aim of our study is to investigate if more patients with hip fracture experience lasting preoperative analgesia until the time of operation or 20 hours after a femoral nerve block with the addition of Dexamethasone compared to the same nerve block done without Dexamethasone.

DETAILED DESCRIPTION:
Patients with hip fractures are most often old, have multiple comorbidities and suffer severe pain.

Femoral nerve block as a means of preoperative analgesia for these patients has proven effective in multiple trials for the majority of the patients. Still some issues remains to be investigated in order to optimize the preoperative analgesia for this group.

One of the issues that reduces the feasibility of the femoral nerve block is the relatively shorter analgesic duration of the nerve block compared to the often longer time from the hospital admission to the actual operation. From the literature and our own experience the mean analgesic duration of a femoral nerve block approximates 15 hours.

Many studies have shown a prolonged analgesic duration of different nerve blocks when Dexamethasone was added to the local anesthetics. Some studies show a 100 percent increase in duration.

To our knowledge no studies have been published regarding prolongation of the analgesic effect of the femoral nerve block with Dexamethasone, and also none regarding the group of patients with hip fracture.

The clinical impact of a femoral nerve block with an analgesic duration of 20 hours compared to the present 15 hours would be less patients waking up in wards during the night time with pain and a terminated femoral nerve block.

The purpose of this study is to investigate if more patients with hip fracture experience a lasting preoperative analgesic duration of at least 20 hours or until the time of operation after a femoral nerve block with Bupivacaine with adrenaline and the addition of Dexamethasone compared to the same nerve block done with only Bupivacaine with adrenaline.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of hip fracture
* Age ≥ 55 years
* Mentally capable of comprehending and using verbal pain score
* Mentally capable of differentiating between pain from the fractured hip and pain from other locations
* Mentally capable of understanding the given information
* Arrival in the emergency room at times when one of the doctors who do the nerve blocks for this investigation are on call
* Verbal pain score (0-10) ≥ 7 with passive leg raise of the fractured leg at the time of inclusion
* Patients informed consent

Exclusion Criteria:

* Hip fracture not confirmed by x-ray
* Weight < 40 kg
* Verbal pain score > 3, 30 minutes after the nerve block
* Verbal pain score > 5 with passive leg raise, 30 minutes after the nerve block
* Patient has previously been included in this trial
* Ongoing pre traumatic treatment with parenteral or intravenous adrenocortical hormone
* Verbal pain score > 3 from other locations than the fractured hip
* If the patient wishes to be excluded
* Allergy to local anesthetics or adrenocortical hormone
* Visible infection in the area of the point of needle injection
* Acute inability to comprehend and use verbal pain score

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Frequency of analgesia at the time of operation or at 20 hours | Until the start of the operation or at 20 hours, average 18 hours
  Frequency of analgesia at the time of operation or at 20 hours in patients with hip fracture after femoral nerve block with Dexamethasone added to Bupivacaine compared to plain Bupivacaine

SECONDARY OUTCOMES:
Frequency of analgesia at the time of operation or at 22 hours | Until the start of the operation or at 22 hours, average 20 hours
  Frequency of analgesia at the time of operation or at 22 hours in patients with hip fracture after femoral nerve block with Dexamethasone added to Bupivacaine compared to plain Bupivacaine
Frequency of analgesia at the time of operation or at 24 hours | Until the start of the operation or at 24 hours, average 22 hours
  Frequency of analgesia at the time of operation or at 24 hours in patients with hip fracture after femoral nerve block with Dexamethasone added to Bupivacaine compared to plain Bupivacaine
Frequency of satisfactory analgesia | Until the start of the operation or at 20 hours, average 18 hours
  Frequency of patients with satisfactory analgesia i the period from the nerve block until the time of operation or at 20 hours compared between the groups
Time to wish for opioid analgesia | Until the start of the operation or at 24 hours, average 22 hours
  Mean time fra nerve block to wish for opioid analgesia compared between groups
Use of opioid analgesia until 20 hours | Until the start of the operation or at 20 hours, average 18 hours
  Mean use of opioid analgesia until the time of operation or at 20 hours compared between groups
Use of opioid analgesia until 22 hours | Until the start of the operation or at 22 hours, average 20 hours
  Mean use of opioid analgesia until the time of operation or at 22 hours compared between groups
Use of opioid analgesia until 24 hours | Until the start of the operation or at 24 hours, average 22 hours
  Mean use of opioid analgesia until the time of operation or at 24 hours compared between groups
Time to analgesic effect with patient at rest | 30 minutes
  Mean time from nerve block to verbal pain score ≤3 at rest
Time to analgesic effect measured while doing passive leg raise | 30 minutes
  Mean time from nerve block to verbal pain score ≤5 while doing passive leg raise
Frequency of insufficient analgesia | 30 minutes
  Frequency of patients with hip fracture with insufficient analgesia after femoral nerve block at 30 minutes
Frequency of absent analgesia | 30 minutes
  Frequency of patients with hip fracture with absent analgesia after femoral nerve block at 30 minutes
Frequency of patients without sufficient analgesia | 30 minutes
  Frequency of patients with hip fracture without sufficient analgesia after femoral nerve block at 30 minutes
Skin sensation in saphenous area | 30 minutes
  Frequency of reduced cold sensation in the skin area innervated by the saphenous nerve when sufficient analgesia versus insufficient analgesia of the fractured hip is experienced 30 minutes after the femoral nerve block
Skin sensation in area of the anterior cutaneous branches of the femoral nerve | 30 minutes
  Frequency of reduced cold sensation in the skin area innervated by the anterior cutaneous branches of the femoral nerve when sufficient analgesia versus insufficient analgesia of the fractured hip is experienced 30 minutes after the femoral nerve block
Sufficient analgesia Dexamethasone vs. plain | 30 minutes
  Success rate of sufficient analgesia after femoral nerve block with Dexamethasone added to Bupivacaine compared to plain bupivacaine
Nerve visualization | Just before injection, which is within an expected average of 10 minutes after inclusion
  Frequency of possible ultrasound visualization of the femoral nerve

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Bendtsen, MD, Ph.d., Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043